CLINICAL TRIAL: NCT04817670
Title: A Phase 2a, Double-blind, Randomised, Placebo-controlled, Efficacy, and Safety Study of Multiple Doses of VIT-2763 in Subjects With Sickle Cell Disease (ViSionSerenity)
Brief Title: Study to Assess Efficacy and Safety of VIT-2763 (Vamifeport) in Subjects With Sickle Cell Disease
Acronym: ViSionSerenity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vifor (International) Inc. (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIT-2763-SCD-202; 2020-005072-34 (EudraCT Number)
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease
Keywords: anemia; sickle cell disease; vamifeport
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia | interventions — VIT-2763

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Participants receive VIT-2763 60 mg, twice a day during 8 weeks.
  Interventions: Drug: VIT-2763 120 mg
- Cohort 2 (Experimental): Participants receive VIT-2763 120 mg, twice a day during 8 weeks.
  Interventions: Drug: VIT-2763 240 mg
- Cohort 3 (Experimental): Participants receive VIT-2763 120 mg, three times a day during 8 weeks.
  Interventions: Drug: VIT-2763 360 mg
- Cohort 4a (Placebo Comparator): Participants receive a placebo, twice a day during 8 weeks.
  Interventions: Drug: Placebo BID
- Cohort 4b (Placebo Comparator): Participants receive a placebo, three times a day during 8 weeks.
  Interventions: Drug: Placebo TID

INTERVENTIONS:
Drug: VIT-2763 120 mg — Participants receive 2 capsules of VIT-2763 30 mg in the morning and in the evening, for 8 weeks.
  Capsules are to be taken orally.
  Other Names: Vamifeport
  Arms: Cohort 1
Drug: VIT-2763 360 mg — Participants receive 2 capsules of VIT-2763 60 mg in the morning, in the afternoon and in the evening for 8 weeks.
  Capsules are to be taken orally.
  Other Names: Vamifeport
  Arms: Cohort 3
Drug: VIT-2763 240 mg — Participants receive 2 capsules of VIT-2763 60 mg in the morning and in the evening, for 8 weeks.
  Capsules are to be taken orally.
  Other Names: Vamifeport
  Arms: Cohort 2
Drug: Placebo BID — Participants receive 2 capsules of placebo in the morning and in the evening, for 8 weeks.
  Capsules are to be taken orally.
  Arms: Cohort 4a
Drug: Placebo TID — Participants receive 2 capsules of Placebo in the morning, in the afternoon and in the evening, for 8 weeks.
  Capsules are to be taken orally.
  Arms: Cohort 4b

SUMMARY:
The purpose of this study is to investigate the effect of VIT-2763 on markers of hemolysis (breakdown in red blood cells) in sickle cell disease (SCD). The safety, tolerability and clinical beneficial effects of VIT-2763 for the treatment of SCD are also explored.

DETAILED DESCRIPTION:
At randomization/baseline, participants are randomized into 3 VIT-2763 dose groups to receive either 60 mg twice daily (BID) (Cohort 1), or 120 mg BID (Cohort 2), or 120 mg 3 times daily (TID) (Cohort 3) and 2 placebo groups (BID, Cohort 4a or TID, Cohort 4b).

The expected duration of patient participation is a maximum of 16 weeks, including a non-treatment screening period of up to 4 weeks, and 8-week treatment period, and a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with confirmed diagnosis of SCD, including only HbS/S or HbS/βT0 genotype.
* Subjects who had at least 1 and no more than 10 vaso-occlusive crises (VOC) episodes reported within 12 months prior to screening.
* Body weight ≥40 kg and ≤120 kg at screening and baseline.
* Subjects on concomitant hydroxyurea must be on a stable dose (mg/kg) for ≥3 months prior to screening Visit V1
* Female subjects of childbearing potential, must have negative pregnancy, must have stopped breastfeeding as of first dose, and must either commit to true abstinence from heterosexual contact or must be willing to use adequate contraceptive precautions.
* Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential

Exclusion Criteria:

* Hb level <6.0 g/dl or >10.4 g/dl for female participants and >11.0 g/dl for male participants, at screening Visit V1
* Having received red blood cell (RBC) transfusion therapy within 4 weeks prior to screening, or ongoing or planned RBC transfusion therapy during the course of the study
* Low levels of Ferritin or transferrin saturation or total iron-binding capacity at screening
* Subjects being hospitalized for SCD-related events within 14 days before the screening visit
* Chronic liver disease or history of liver cirrhosis, and/or high levels of alanine aminotransferase or aspartate aminotransferase at baseline
* Low estimated glomerular filtration rate, and/or significant high urinary albumin/creatinine ratio at screening or on chronic dialysis.
* Newly diagnosed folate deficiency anemia, which is considered clinically relevant by the Investigator at screening
* Any history or clinically important finding of cardiac or pulmonary disorders
* Family history of long-QT syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death
* Clinically significant bacterial, fungal, parasitic, or viral infection which requires therapy. Note: A subject meeting this criterion should delay screening and/or enrolment for a minimum of 2 weeks, or if excluded can be re-screened at a later time point.
* Concomitant use of certain hormonal contraceptives as defined in the study protocol, are not allowed within 4 weeks prior to screening and until 1 week after the last administration of the study drug and the use of progesterone-only hormonal contraception as the sole measure to prevent pregnancy.
* Pregnant or females currently breastfeeding.
* History or known concomitant solid tumours and/or haematological malignancies unless resolved in the ≥2 past years, except for basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, incidental histologic finding of prostate cancer
* Unable to take and absorb oral medications
* Acute peptic stomach or duodenal ulcer in the previous 6 months before screening and/or healed after 3 months of treatment.
* Uncontrolled hemorrhages

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Hermosilla, PhD, Study Director — Vifor (International) Inc.
Locations (22):
- United States (8):
  - Investigator Site 709, Birmingham, Alabama
  - Investigator Site 708, Los Angeles, California
  - Investigator Site 713, Aurora, Colorado
  - Investigator Site 706, Hollywood, Florida
  - Investigator Site 703, Chicago, Illinois
  - Investigator Site 701, Greenville, North Carolina
  - Investigator Site 711, Charleston, South Carolina
  - Investigator Site 702, Milwaukee, Wisconsin
- France (2):
  - Investigator Site 801, Colombes
  - Investigator Site 802, Lyon
- Greece (3):
  - Investigator Site 305, Athens
  - Investigator site 301, Athens
  - Investigator Site 302, Pátrai
- Lebanon (3):
  - Investigator Site 101, Baabda
  - Investigator Site 102, Beirut
  - Investigator Site 103, Tripoli
- United Kingdom (6):
  - Investigator Site 606, Liverpool
  - Investigator Site 603, London
  - Investigator Site 608, London
  - Investigator Site 601, London
  - Investigator Site 605, London
  - Investigator Site 607, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nyffenegger N, Zennadi R, Kalleda N, Flace A, Ingoglia G, Buzzi RM, Doucerain C, Buehler PW, Schaer DJ, Durrenberger F, Manolova V. The oral ferroportin inhibitor vamifeport improves hemodynamics in a mouse model of sickle cell disease. Blood. 2022 Aug 18;140(7):769-781. doi: 10.1182/blood.2021014716. PMID 35714304
- [Derived] Parrow NL, Doherty JM, Conrey A, Thein SL, Fleming RE. Relationships Between Markers of Iron Status and Hematological Parameters in Patients With Sickle Cell Disease. Adv Hematol. 2024 Dec 3;2024:9872440. doi: 10.1155/ah/9872440. eCollection 2024. PMID 39659429
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35714304/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 22 sites initiated for this study in 5 countries (The United Kingdom, Lebanon, Greece, the United States, and France).
Pre-assignment Details: A total of 46 participants were screened in this study, of which 28 were screen failures. Out of these 28 participants, 9 were rescreened, and 7 were found eligible for the study. 25 participants were enrolled in the study.
Groups:
- Cohort 1: VIT-2763 60 mg BID (120 mg/Day): Participants received VIT-2763 60 milligrams (mg) (2 x 30 mg capsules), orally, twice daily (BID) for 8 weeks.
- Cohort 2: VIT-2763 120 mg BID (240 mg/Day): Participants received VIT-2763 120 mg (2 x 60 mg capsules), orally, BID for 8 weeks.
- Cohort 3: VIT-2763 120 mg TID (360 mg/Day): Participants received VIT-2763 120 mg (2 x 60 mg capsules), orally, three times daily (TID) for 8 weeks.
- Cohort 4: Placebo: Participants received placebo capsules, orally, BID or TID for 8 weeks.
- Cohort 2a: VIT-2763 30 mg BID (60 mg/Day): One participant received VIT-2763 30 mg, orally, BID for 8 weeks under Protocol Version 2.0. However, after the implementation of Protocol Version 3.0 and higher, this participant was excluded from the efficacy analysis and only safety data were reported (as planned).
Period: Overall Study
Arm/Group | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) | Cohort 4: Placebo | Cohort 2a: VIT-2763 30 mg BID (60 mg/Day)
Started | 6 | 6 | 6 | 6 | 1
Intent-to-treat (ITT) Population (The ITT population consisted of all participants who were randomly assigned to a treatment group.) | 6 | 6 | 6 | 6 | 0
Completed | 5 | 6 | 5 | 6 | 1
Not Completed | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis was performed on the safety set. The safety set consisted of all randomized participants who had taken at least one dose of investigational medicinal product (IMP). Data for Cohort 2a are not reported here because of concerns regarding participant privacy as there was only 1 participant in the Cohort 2a arm.
Groups:
- Cohort 1: VIT-2763 60 mg BID (120 mg/Day): Participants received VIT-2763 60 mg (2 x 30 mg capsules), orally, BID for 8 weeks.
- Cohort 3: VIT-2763 120 mg TID (360 mg/Day): Participants received VIT-2763 120 mg (2 x 60 mg capsules), orally, TID for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) | Cohort 4: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (7.41) | 36.0 (11.87) | 29.3 (9.48) | 25.3 (7.17) | 30.2 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 3 | 13
  Male | 2 | 3 | 3 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 5 | 6 | 22
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 3 | 4 | 12
  White | 4 | 3 | 2 | 2 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Haemolysis Marker (Indirect Bilirubin)
Description: Mean change from baseline in haemolysis markers was measured by reduction of indirect bilirubin.
Time Frame: Baseline and after 8 weeks of treatment
Population: This analysis was performed on the intent-to-treat (ITT) population. The ITT population consisted of all participants who were randomly assigned to a treatment group under Protocol Version 3.0 or higher. Here, the 'overall number of participants analyzed' (N) signifies the number of participants with evaluable data for this outcome measure. The 'number analyzed' (n) signifies the number of participants with evaluable data for each specified timepoint.
Measure: Mean (Standard Deviation); unit: micromoles per liter (umol/L)
Arm/Group | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) | Cohort 4: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 6
micromoles per liter (umol/L)
  Baseline | 24.0 (13.51) | 56.4 (43.71) | 44.0 (24.48) | 31.2 (12.95)
  Change at 8 weeks: number analyzed (Participants) | 4 | 4 | 4 | 5
  Change at 8 weeks | -4.0 (4.69) | -5.8 (11.35) | -21.8 (11.62) | 0.6 (7.30)

2. Secondary Outcome: Mean Change From Baseline in Haemolysis Marker (Direct and Total Bilirubin)
Description: Mean change from baseline in haemolysis markers was measured by direct and total bilirubin.
Time Frame: Baseline and after 8 weeks of treatment
Population: This analysis was performed on the ITT population. The ITT population consisted of all participants who were randomly assigned to a treatment group under Protocol Version 3.0 or higher. Here, the 'overall number of participants analyzed' (N) signifies the number of participants with evaluable data for this outcome measure. The 'number analyzed' (n) signifies the number of participants with evaluable data for each specified category.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) | Cohort 4: Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 6
umol/L
  Direct Bilirubin: number analyzed (Participants) | 4 | 4 | 4 | 5
  Direct Bilirubin | -0.5 (1.29) | -2.0 (2.83) | -2.5 (7.05) | -0.4 (1.52)
  Total Bilirubin | -4.2 (4.76) | -13.2 (16.57) | -26.0 (16.00) | -0.2 (7.08)

3. Secondary Outcome: Mean Change From Baseline in Haemolysis Marker (Lactate Dehydrogenase)
Description: Mean change from baseline in haemolysis markers was measured by lactate dehydrogenase.
Time Frame: Baseline and after 8 weeks of treatment
Population: This analysis was performed on the ITT population. The ITT population consisted of all participants who were randomly assigned to a treatment group under Protocol Version 3.0 or higher. Here, the 'overall number of participants analyzed' (N) signifies the number of participants with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) | Cohort 4: Placebo
Number analyzed (Participants) | 4 | 3 | 3 | 5
units per liter (U/L) | -45.8 (47.56) | -24.0 (6.08) | 7.7 (197.50) | 47.8 (60.06)

4. Secondary Outcome: Mean Change From Baseline in Haemolysis Marker (Potassium)
Description: Mean change from baseline in haemolysis markers was measured by potassium.
Time Frame: Baseline and after 8 weeks of treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) | Cohort 4: Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 6
millimoles per liter (mmol/L) | 0.08 (0.396) | 0.08 (0.192) | -0.22 (0.319) | -0.05 (0.295)

5. Secondary Outcome: Mean Change From Baseline in Haemolysis Marker (Hemoglobin and Haptoglobin)
Description: Mean change from baseline in haemolysis markers was measured by hemoglobin and haptoglobin.
Time Frame: Baseline and after 8 weeks of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) | Cohort 4: Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 6
grams per liter (g/L)
  Hemoglobin: number analyzed (Participants) | 5 | 6 | 4 | 6
  Hemoglobin | -3.400 (1.4748) | -2.067 (5.5142) | -1.575 (8.4017) | 2.733 (9.9933)
  Haptoglobin | 0.102 (0.2281) | -0.012 (0.0286) | 0.528 (0.8312) | 0.000 (0.0000)

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), TEAEs Related to IMP and by Severity of TEAEs
Description: TEAEs were defined as adverse events (AEs) with an onset date later or on the same date as first investigational medicinal product (IMP) intake. The severity grading was determined according to the Common Terminology Criteria for AEs, where the Common Terminology Criteria grades relate to severity as follows: Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-threatening and Grade 5: Death.
Time Frame: From first dose of study drug up to 12 weeks
Population: Analysis was performed on the safety set. The safety set consists of all randomized participants (under Protocol Version 3.0 or higher) who had taken at least one dose of IMP. The participants in the safety set were analyzed based on the treatment they received, regardless of randomization. Data are separately reported for the one participant in the Cohort 2a arm (randomized under Protocol Version 2.0).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) | Cohort 4: Placebo | Cohort 2a: VIT-2763 30 mg BID (60 mg/Day)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 1
Participants
  Any TEAEs | 4 | 4 | 5 | 5 | 1
  TEAEs related to IMP | 0 | 0 | 0 | 1 | 0
  TEAEs with severity: Mild | 0 | 3 | 2 | 3 | 1
  TEAEs with severity: Moderate | 3 | 1 | 1 | 2 | 1
  TEAEs with severity: Severe | 1 | 0 | 2 | 0 | 0
  TEAEs with severity: Life threatening | 0 | 0 | 0 | 0 | 0
  TEAEs with severity: Death | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 12 weeks
Description: Analysis was performed on the safety set. The safety set consists of all randomized participants (under Protocol Version 3.0 or higher) who had taken at least one dose of IMP. The participants in the safety set were analyzed based on the treatment they received, regardless of randomization. Data are separately reported for the one participant in the Cohort 2a arm (randomized under Protocol Version 2.0).
Arm/Group | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) | Cohort 4: Placebo | Cohort 2a: VIT-2763 30 mg BID (60 mg/Day)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 1/6 | 1/1
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 5/6 | 5/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) (N=6) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) (N=6) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) (N=6) | Cohort 4: Placebo (N=6) | Cohort 2a: VIT-2763 30 mg BID (60 mg/Day) (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: VIT-2763 60 mg BID (120 mg/Day) (N=6) | Cohort 2: VIT-2763 120 mg BID (240 mg/Day) (N=6) | Cohort 3: VIT-2763 120 mg TID (360 mg/Day) (N=6) | Cohort 4: Placebo (N=6) | Cohort 2a: VIT-2763 30 mg BID (60 mg/Day) (N=1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 3 | 1 | 2 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0
Sickle cell disease (Congenital, familial and genetic disorders) | 0 | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pallor (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT04817670/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT04817670/SAP_001.pdf